CLINICAL TRIAL: NCT01515436
Title: A Randomized, Single-Blinded Clinical Trial: The Effect of Music Periodicity on Interictal Epileptiform Discharges
Brief Title: The Effect of Music Periodicity on Interictal Epileptiform Discharges
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Robert P. Turner, Dr. Robert Turner, Medical University of South Carolina
Allocation: Randomized | Masking: Single | Purpose: Treatment
Other Study IDs: HR11247
Record Dates: First submitted 2012-01-18; First posted 2012-01-24 (Estimated); Last update posted 2012-01-24 (Estimated); Status verified 2012-01

CONDITIONS: Rolandic Epilepsy; Benign Childhood Epilepsy With Centrotemporal Spikes; Epilepsy; Seizures
Keywords: Rolandic Epilepsy; Benign Childhood Epilepsy with Centrotemporal Spikes (BCECTS); Epilepsy; Seizures; Music; Mozart; Beethoven
MeSH Terms: conditions — Epilepsy, Rolandic; Epilepsy; Seizures

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mozart alternating with Beethoven (Active Comparator): Study participants will listen to Mozart's Sonata for Two Pianos in D Major, K. 448 alternating with Beethoven's Fur Elise.
  Interventions: Other: Mozart alternating with Beethoven
- Beethoven alternating with Mozart (Active Comparator): Study participants will listen to Beethoven's Fur Elise alternating with Mozart's Sonata for Two Pianos in D Major, K. 448.
  Interventions: Other: Beethoven alternating with Mozart

INTERVENTIONS:
Other: Mozart alternating with Beethoven — Study participants will listen to Mozart's Sonata for Two Pianos in D Major, K. 448 alternating with Beethoven's Fur Elise.
  Arms: Mozart alternating with Beethoven
Other: Beethoven alternating with Mozart — Study participants will listen to Beethoven's Fur Elise alternating with Mozart's Sonata for Two Pianos in D Major, K. 448.
  Arms: Beethoven alternating with Mozart

SUMMARY:
The purpose of this study is to determine if having children listen to the music of Wolfgang Amadeus Mozart (Sonata for Two Pianos in D Major, K. 448) will lessen the amount of spike discharges on his/her Electroencephalography (EEG). These spike discharges often occur during a 24 hour period in the EEG of a child with Benign Childhood Epilepsy with Centrotemporal Spikes (BCECTS), or Rolandic Epilepsy. Should there be a decrease in the amount of spike discharges after listening to Mozart's music, this information may lead to new understanding and possible treatments for epilepsy.

ELIGIBILITY:
Inclusion Criteria:

* Female or male with BCECTS clinical history, and at least one seizure, as defined by the International League Against Epilepsy.
* EEG consistent with features of BCECTS: centrotemporal (rolandic) interictal spike discharges (ISDs) with otherwise normal background interictal EEG
* Screening neurological examination normal (by PI or other pediatric neurologist in the Division of Pediatric Neurology at MUSC)
* Age 5-12 years, inclusive
* On less than or equal to 2 anti-epileptic drugs (AED) [Range 0-2 AEDs]

Exclusion Criteria:

* Currently taking Clonazepam or other Benzodiazepines
* Inability to complete 12 hour admission and comply with study protocol
* Prohibited Therapy or Activities During Study Period: Use of computer or video games. Viewing of video tapes will be prohibited due to potential effect of music in videos on underlying process of study.
* Due to the confounding factor of probably suppression of IEDs after a clinical seizure, any subject experiencing a seizure of any duration 24 hours prior to beginning the study will be excluded from the study.
* For any subject experiencing a seizure during the study, data analysis will cease from that point onward.

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2004-02; Primary Completion 2004-05 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert P Turner, MD, MSCR, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States